CLINICAL TRIAL: NCT05738564
Title: Pre-emptive Epinephrine Nebulization Prior to Nasotracheal Intubation for Mandibular Fracture Fixation Surgeries:Dose it Really Differs? a Randomized Controlled Study
Brief Title: Epinephrine Nebulization Prior to Nasotracheal Intubation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: FMASU R 132/2021
Record Dates: First submitted 2023-01-11; First posted 2023-02-22 (Actual); Last update posted 2023-02-22 (Actual); Status verified 2023-02

CONDITIONS: Nasal Bleeding
Keywords: Nasotracheal intubation, nebulized epinephrine, epistaxis.
MeSH Terms: conditions — Epistaxis

STUDY DESIGN:
Intervention Model Description: Randomised, prospective trial performed on 2 equal groups
Who Masked: Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group (EL) Epinepherine and Lidocaone group (Active Comparator): Group (EL) (63 patients) received a session of nebulization in the pre-induction area, consisting of 1 ml epinephrine (1:1000 Martindale Pharma, an Ethypharm Group Company, ampoule 1 mg added to 9 ml of normal saline, then 1 ml of that put in nebulization cup + 2 ml lidocaine 2%), nebulized prior to the induction of anesthesia.(63 patients) received a session of nebulization in the pre-induction area, consisting of 1 ml epinephrine (1:1000 Martindale Pharma, an Ethypharm Group Company, ampoule 1 mg added to 9 ml of normal saline, then 1 ml of that put in nebulization cup + 2 ml lidocaine 2%), nebulized prior to the induction of anesthesia.
  Interventions: Drug: Epinephrine Inhalation Solution
- Group( OL) Oxymetazoline and lidocaine group (Active Comparator): Group OL (63 patients): These patients received five drops of lidocaine hydrochloride (Xylocaine 2%, 20 mg/ml; AstraZeneca, London, UK) using a prefilled dropper, followed by six drops of hydrochloride Oxymetazoline (Otrivin adult nasal drops 0.1%, 10 ml of 1 mg/ml; Novartis Consumer Health, UK Ltd, 980 Great West Road, Brentford, Middlesex, TW8 9GS, UK) in each nostril in the pre-induction room just before the induction of anesthesia
  Interventions: Drug: Epinephrine Inhalation Solution

INTERVENTIONS:
Drug: Epinephrine Inhalation Solution — epinephrine prepared solution mixed with lidocaine (EL) Otrivin adult nasal drops 0.1Otrivin adult nasal drops 0.1%, 10 ml of 1 mg/ml; Novartis Consumer Health, UK Ltd, 980 Great West Road, Brentford, Middlesex, TW8 9GS, UK) in each nostril in the pre-induction room just before the induction of anesthesia
  Other Names: oxymetazoline lidocaine

SUMMARY:
This randomised, prospective study performed in Ain shams university hospitals over 126 Patients ASA I and ASA II, trauma patients who suffered isolated mandibular fractures and necessitated nasal intubation during general anesthesia. The patients were randomly assigned to one of two equal groups: nasal Lidocaine drops followed by Oxymetazoline nasal drops group (OL) or Epinephrine mixed with Lidocaine as nebulization session (EL) group.

DETAILED DESCRIPTION:
One group received epinephrine mixed with lidocaine as nebulization session (EL group) and the other group received nasal lidocaine drops followed by Oxymetazoline nasal drops group (OL). Before the preparation of the airway, we examined the nasal cavity by using a light source to select the target nostril; if we could not determine, we chose the right nostril. No premedication was administered.

Group (EL) (63 patients) received a session of nebulization in the pre-induction area, consisting of 1 ml epinephrine (1:1000 Martindale Pharma, an Ethypharm Group Company, ampoule 1 mg added to 9 ml of normal saline, then 1 ml of that put in nebulization cup + 2 ml lidocaine 2%), nebulized prior to the induction of anesthesia.

Group OL (63 patients): These patients received five drops of lidocaine hydrochloride (Xylocaine 2%, 20 mg/ml; AstraZeneca, London, UK) using a prefilled dropper, followed by six drops of hydrochloride Oxymetazoline (Otrivin adult nasal drops 0.1%, 10 ml of 1 mg/ml; Novartis Consumer Health, UK Ltd, 980 Great West Road, Brentford, Middlesex, TW8 9GS, UK) in each nostril in the

ELIGIBILITY:
Inclusion Criteria:

* Cases with American Society of Anesthesiologists (ASA) classes I and II.
* Patients scheduled for elective oral isolated mandibular fracture fixation requiring nasotracheal intubation.

Exclusion Criteria:

* Nasal abnormality history (such as polyp , surgery or nasal trauma).
* Frequent epistaxis history.
* Patients suffering valvular heart disease, hypertension, ischemic heart disease or arrhythmias.
* Patients using drugs (anticoagulation therapy, non-steroidal anti-inflammatory drugs, and oral decongestants).
* Patients receiving medications known to alter the parameters under investigation including β-blockers, calcium channel blockers, or vasodilators.
* Patients known to have hypersensitivity to medications used in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
estimate the degree of epistaxis | the whole intraoperative time
  Epistaxis degrees during intubation is classified to 4 degrees 1-No bleeding means No interference with the laryngoscopic view,2- minimal bleeding means Just blood-tinged ETT but no blood on the vocal cords or mouth floor, 3-moderate bleading means Blood on the vocal cords and mouth floor which Interferes with the laryngoscopic view, but is easy to confirm the laryngeal structure,4-severe bleeding means Blood on the vocal cords and mouth floor Hard to visualize the laryngeal structure without suction because of bleeding Nasal bleeding after intubation will be assessed by utilizing pharyngeal aspiration with a 14-F, 50-cm-long suction catheter linked to a 2.5-m-long suction tube at -100 mmHg pressure [13]. Based on the amount of blood sucked via the suction tube into the container, the severity of epistaxis was determined: none = no bleeding; mild = blood volume < 50 cm; moderate = 50 cm < blood volume < 300 cm; severe = blood volume > 300 cm

SECONDARY OUTCOMES:
intraoperative analgesia | the whole intraoperative period
  intraoperative analgesia is indicated by intraoperative hemodynamics and total intraoperative fentanyl consumption
intraoperative blood loss from surgical field | the whole intraoperative period
  itraoperative volume of blood loss was estimated

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed Shorbagy, MD, Principal Investigator — Assisstant professor of anesthesia
Locations (1):
- Ain Shams University Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
through the official email
Supporting Information: Study Protocol, CSR
Time Frame: after 1 month will be available for 6 months
Access Criteria: through the official email sabah_nageeb@med.asu.edu.eg

REFERENCES:
- [Background] Song J. A comparison of the effects of epinephrine and xylometazoline in decreasing nasal bleeding during nasotracheal intubation. J Dent Anesth Pain Med. 2017 Dec;17(4):281-287. doi: 10.17245/jdapm.2017.17.4.281. Epub 2017 Dec 28. PMID 29349350